CLINICAL TRIAL: NCT04594239
Title: Evaluation of Effectiveness and Safety of Belotero Balance® (+) Lidocaine for Volume Augmentation of the Infraorbital Hollow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M930121002
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Volume Loss in the Infraorbital Hollow Area
MeSH Terms: interventions — Needles; Cannula; Treatment Delay

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Treatment, needle (Experimental)
  Interventions: Device: Belotero Balance (+) Lidocaine, needle
- Treatment, cannula (Experimental)
  Interventions: Device: Belotero Balance (+) Lidocaine, cannula
- Untreated-control / delayed-treatment, needle (Other)
  Interventions: Device: Untreated-control / delayed-treatment, needle
- Untreated-control / delayed-treatment, cannula (Other)
  Interventions: Device: Untreated-control / delayed-treatment, cannulas

INTERVENTIONS:
Device: Belotero Balance (+) Lidocaine, needle — Injection of Belotero Balance (+) Lidocaine to the infraorbital hollows using needles
  Arms: Treatment, needle
Device: Belotero Balance (+) Lidocaine, cannula — Injection of Belotero Balance (+) Lidocaine into the infraorbital hollows using cannulas
  Arms: Treatment, cannula
Device: Untreated-control / delayed-treatment, needle — Untreated-control, followed by delayed-treatment with Belotero Balance (+) Lidocaine (injection of Belotero Balance (+) Lidocaine to the infraorbital hollows using needles)
  Arms: Untreated-control / delayed-treatment, needle
Device: Untreated-control / delayed-treatment, cannulas — Untreated-control, followed by delayed-treatment with Belotero Balance (+) Lidocaine (injection of Belotero Balance (+) Lidocaine to the infraorbital hollows using cannulas)
  Arms: Untreated-control / delayed-treatment, cannula

SUMMARY:
* Confirm the effectiveness of Belotero Balance® (+) Lidocaine (BBL) injection for the correction of volume loss in the infraorbital hollow (IOH) area by demonstrating superiority to untreated control.
* Confirm the safety of BBL injection for the correction of volume loss in the IOH area.

ELIGIBILITY:
Inclusion Criteria:

* Is a candidate for bilateral IOH treatment.
* Has symmetrical right and left IOHs with the same MIHAS score of 2 or 3 (moderate or severe), as assessed live by the blinded evaluator.

Exclusion Criteria:

* Prior lower-eyelid surgery, including orbital or midface surgery, or a permanent implant or graft in the midfacial region that could interfere with effectiveness assessments.
* Previous treatment with fat injections or permanent and/or semi-permanent dermal fillers in the midfacial region.
* Previous lower-eyelid and/or malar-region treatments with any dermal fillers (e.g., collagen, hyaluronic acid (HA), calcium hydroxyapatite, poly L-lactic acid (PLLA)) within the past 24 months.
* Any other medical condition with the potential to interfere with the study outcome assessments or compromise subject safety.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (9):
- United States (8):
  - Art of Skin MD, Merz Investigational Site #0010444, Solana Beach, California
  - Moradi MD Face Beautiful Inc., Merz Investigational Site #0010358, Vista, California
  - MetroDerm / Atlanta Center for Clinical Research, Merz Investigational Site #0010446, Atlanta, Georgia
  - Project Glammers, Merz Investigational Site #0010443, Brooklyn, New York
  - The Center for Dermatology, Cosmetic & Laser Surgery, Merz Investigational Site #0010442, Mount Kisco, New York
  - Mariwalla Dermatology, Merz Investigational Site #0010445, West Islip, New York
  - HKB Surgeons, Merz Investigational Site #0010447, Huntersville, North Carolina
  - Nashville Centre for Laser & Facial Surgery, Merz Investigational Site #0010353, Nashville, Tennessee
- Jose Raul Montes Eyes and Facial Rejuvenation, Merz Investigational Site #0010436, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 9 investigational sites in the United States.
Pre-assignment Details: Of the 187 screened subjects, 37 were exited as screen failures.150 subjects were enrolled and randomized in this study.
Groups:
- Belotero Balance (+) Lidocaine (BBL) Treatment With Needle: Subjects received a single treatment of BBL injection using needle in both infraorbital hollow (IOH) areas at Day 1 and 48 weeks after last injection (optional retreatment). Subjects were eligible to receive an optional touch-up injection 4 weeks after initial injection.
- BBL Treatment With Cannula: Subjects received a single treatment of BBL injection using cannula in both IOH areas at Day 1 and 48 weeks after last injection (optional retreatment). Subjects were eligible to receive an optional touch-up injection 4 weeks after initial injection.
- Control/Delayed-treatment BBL With Needle: Subjects were untreated until Week 8 and then received a single treatment of BBL injection using needle in both IOH areas. Subjects were eligible to receive an optional touch-up injection 4 weeks after initial injection.
- Control/Delayed-treatment BBL With Cannula: Subjects were untreated until Week 8 and then received a single treatment of BBL injection using cannula in both IOH areas. Subjects were eligible to receive an optional touch-up injection 4 weeks after initial injection.
Period: Overall Study
Arm/Group | Belotero Balance (+) Lidocaine (BBL) Treatment With Needle | BBL Treatment With Cannula | Control/Delayed-treatment BBL With Needle | Control/Delayed-treatment BBL With Cannula
Started | 49 | 48 | 27 | 26
Safety Population | 49 | 48 | 26 | 21
Completed | 38 | 39 | 21 | 15
Not Completed | 11 | 9 | 6 | 11
Not completed — Withdrawal by Subject | 3 | 4 | 2 | 4
Not completed — Lost to Follow-up | 8 | 5 | 4 | 6
Not completed — Subject relocated | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized and treated subjects of the treatment group as well as all randomized subjects of the control/delayed-treatment groups.
Groups:
- BBL Treatment With Needle: Subjects received a single treatment of BBL injection using needle in both IOH areas at Day 1 and 48 weeks after last injection (optional retreatment). Subjects were eligible to receive an optional touch-up injection 4 weeks after initial injection.
- Total: Total of all reporting groups
Arm/Group | BBL Treatment With Needle | BBL Treatment With Cannula | Control/Delayed-treatment BBL With Needle | Control/Delayed-treatment BBL With Cannula | Total
Number analyzed (Participants) | 49 | 48 | 27 | 26 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (9.06) | 44.3 (9.05) | 43.2 (10.83) | 40.0 (9.18) | 43.3 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 36 | 22 | 23 | 125
  Male | 5 | 12 | 5 | 3 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 16 | 7 | 7 | 50
  Not Hispanic or Latino | 29 | 32 | 20 | 19 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 2
  Black or African American | 3 | 6 | 3 | 5 | 17
  White | 40 | 33 | 19 | 17 | 109
  More than one race | 5 | 5 | 2 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate Based on Merz Infraorbital Hollow Assessment Scale (MIHAS) at Week 8
Description: Responder rate was defined as percentage of subjects with treatment response at Week 8 on MIHAS, as assessed live by a blinded evaluator. Responders were defined as subjects who achieved greater than or equal to (>=) 1 grade improvement on both IOHs on the MIHAS. MIHAS (to assess infraorbital hollow) was a 5-point scale ranging as: Grade 0 (none to minimal), Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (extreme). A higher score indicated extreme signs of hollowing. This analysis was done using multiple imputation method to impute missing MIHAS scores. Percentage of subjects with response at Week 8 and corresponding confidence intervals were average values obtained from the multiple imputation approach.
Time Frame: Week 8
Population: ITT. As planned, the data for this outcome measure was analyzed for pooled BBL treatment groups (needle and cannula), BBL treatment with needle group, BBL treatment with cannula group and pooled control/delayed-treatment groups BBL (needle and cannula).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- BBL Treatment: All Subjects: Subjects received a single treatment of BBL injection using needle and cannula in IOH area at Day 1 and 48 weeks after last injection (optional retreatment). Subjects were eligible to receive an optional touch-up injection 4 weeks after initial injection.
- Control/Delayed-treatment BBL: All Subjects: Subjects were untreated until Week 8 and then received a single treatment of BBL injection using needle and cannula in both IOH areas. Subjects were eligible to receive an optional touch-up injection 4 weeks after initial injection.
Arm/Group | BBL Treatment: All Subjects | BBL Treatment With Needle | BBL Treatment With Cannula | Control/Delayed-treatment BBL: All Subjects
Number analyzed (Participants) | 97 | 49 | 48 | 53
percentage of subjects | 80.6 [71.4 to 87.4] | 87.4 [75.0 to 94.1] | 73.7 [59.4 to 84.3] | 1.9 [0.3 to 10.2]
Statistical Analysis 1: Comparison: BBL Treatment: All Subjects vs Control/Delayed-treatment BBL: All Subjects; Test type: Superiority; Difference in response rates = 78.7, 95% CI 2-sided [66.3 to 85.6]
Statistical Analysis 2: Comparison: BBL Treatment With Needle vs Control/Delayed-treatment BBL: All Subjects; Test type: Superiority; Difference in response rates = 85.4, 95% CI 2-sided [70.5 to 92.3]
Statistical Analysis 3: Comparison: BBL Treatment With Cannula vs Control/Delayed-treatment BBL: All Subjects; Test type: Superiority; Difference in response rates = 71.8, 95% CI 2-sided [55.2 to 82.5]

2. Secondary Outcome: Percentage of Subjects With Global Aesthetic Improvement Scale (GAIS) Score at Week 8, as Assessed by the Treating Investigator
Description: The GAIS is a 7-point scale ranging as +3 (very much improved); +2 (much improved); +1 (improved); 0 (no change); -1 (worse); -2 (much worse); -3 (very much worse), as assessed by the investigator. An improvement on the GAIS was classified as "improved", "much improved", or "very much improved.
Time Frame: Week 8
Population: ITT. Here "overall number of subjects analyzed" were subjects who were evaluable for this outcome measure that is, subjects with observed data. As planned, the data for this outcome measure was calculated and analyzed only for subjects randomized to the treatment groups (needle and cannula).
Measure: Number; unit: percentage of subjects
Arm/Group | BBL Treatment With Needle | BBL Treatment With Cannula
Number analyzed (Participants) | 46 | 43
percentage of subjects
  Very Much Improved (+3) | 47.8 | 44.2
  Much Improved (+2) | 41.3 | 25.6
  Improved (+1) | 8.7 | 30.2
  No Change (0) | 2.2 | 0
  Worse (-1) | 0 | 0
  Much Worse (-2) | 0 | 0
  Very Much Worse (-3) | 0 | 0

3. Secondary Outcome: Percentage of Subjects With GAIS Score at Week 8, as Assessed by the Subject
Description: The GAIS is a 7-point scale ranging as +3 (very much improved); +2 (much improved); +1 (improved); 0 (no change); -1 (worse); -2 (much worse); -3 (very much worse), as assessed by the subject. An improvement on the GAIS was classified as "improved", "much improved", or "very much improved.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | BBL Treatment With Needle | BBL Treatment With Cannula
Number analyzed (Participants) | 46 | 43
percentage of subjects
  Very Much Improved (+3) | 34.8 | 30.2
  Much Improved (+2) | 45.7 | 37.2
  Improved (+1) | 19.6 | 32.6
  No Change (0) | 0 | 0
  Worse (-1) | 0 | 0
  Much Worse (-2) | 0 | 0
  Very Much Worse (-3) | 0 | 0

4. Secondary Outcome: Change From Baseline in Rasch-Transformed Score for the Face-Q Satisfaction With Eyes at Week 8
Description: The FACE-Q is a set of standardized patient-reported outcome scales for subjects undergoing facial cosmetic procedures. Subjects answered 7 questions of the FACE-Q satisfaction with eyes using a 4- point scale where: 1(very dissatisfied), 2 (somewhat dissatisfied), 3 (somewhat satisfied), 4 (very satisfied). The sum FACE-Q scores were Rasch-transformed and ranged from 0 to 100. Higher scores reflected a better outcome (greater satisfaction).
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BBL Treatment With Needle | BBL Treatment With Cannula
Number analyzed (Participants) | 46 | 43
score on a scale | 27.4 (26.0) | 24.6 (27.9)

5. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) Related to BBL
Description: TEAEs are defined as adverse events (AEs) with onset or worsening on or after date and time of first dose of study treatment. A TEAE was considered to be "related" if a causal relationship between BBL and the TEAE is at least reasonably possible.
Time Frame: BBL Treatment (Needle and Cannula): Up to 80 weeks; Control/Delayed-treatment BBL (Needle and Cannula): Up to 56 weeks
Population: The Safety Population (SP) included all treated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | BBL Treatment With Needle | BBL Treatment With Cannula | Control/Delayed-treatment BBL With Needle | Control/Delayed-treatment BBL With Cannula
Number analyzed (Participants) | 49 | 48 | 26 | 21
Participants | 5 | 6 | 1 | 1

6. Secondary Outcome: Number of Subjects With Treatment-Emergent Serious Adverse Events (TESAEs) Related to BBL
Description: TESAEs included TEAEs that resulted in death, required either inpatient hospitalization or the prolongation of hospitalization, were life-threatening, resulted in a persistent or significant disability/incapacity or resulted in a congenital anomaly/birth defect. A TESAE was considered to be "related" if a causal relationship between BBL and the TESAE is at least reasonably possible.
Time Frame: BBL Treatment (Needle and Cannula): Up to 80 weeks; Control/Delayed-treatment BBL (Needle and Cannula): Up to 56 weeks
Population: SP.
Measure: Count of Participants; unit: Participants
Arm/Group | BBL Treatment With Needle | BBL Treatment With Cannula | Control/Delayed-treatment BBL With Needle | Control/Delayed-treatment BBL With Cannula
Number analyzed (Participants) | 49 | 48 | 26 | 21
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: BBL Treatment (Needle and Cannula): Up to 80 weeks; Control/Delayed-treatment BBL (Needle and Cannula): Up to 8 weeks; Delayed-treatment BBL (Needle and Cannula): Up to 48 weeks
Description: The investigator reported adverse events (AEs) systematically at each visit. The data for AEs was reported as per treatment received by the subject.
Groups:
- Control/Delayed-treatment BBL With Needle: Subjects randomized to Delayed-treatment BBL With Needle from randomization until initial treatment at Week 8.
- Delayed-treatment BBL With Needle: Subjects received a single treatment of BBL injection using needle in both IOH areas at Week 8 and were eligible to receive an optional touch-up injection 4 weeks after initial injection.
- Control/Delayed-treatment BBL With Cannula: Subjects randomized to Delayed-treatment BBL With Cannula from randomization until initial treatment at Week 8.
- Delayed-treatment BBL With Cannula: Subjects received a single treatment of BBL injection using cannula in both IOH areas at Week 8 and were eligible to receive an optional touch-up injection 4 weeks after initial injection.
Arm/Group | BBL Treatment With Needle | BBL Treatment With Cannula | Control/Delayed-treatment BBL With Needle | Delayed-treatment BBL With Needle | Control/Delayed-treatment BBL With Cannula | Delayed-treatment BBL With Cannula
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48 | 0/27 | 0/26 | 0/26 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/48 | 0/27 | 0/26 | 0/26 | 0/21
Other Adverse Events (participants affected / at risk) | 6/49 | 11/48 | 0/27 | 4/26 | 0/26 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BBL Treatment With Needle (N=49) | BBL Treatment With Cannula (N=48) | Control/Delayed-treatment BBL With Needle (N=27) | Delayed-treatment BBL With Needle (N=26) | Control/Delayed-treatment BBL With Cannula (N=26) | Delayed-treatment BBL With Cannula (N=21)
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BBL Treatment With Needle (N=49) | BBL Treatment With Cannula (N=48) | Control/Delayed-treatment BBL With Needle (N=27) | Delayed-treatment BBL With Needle (N=26) | Control/Delayed-treatment BBL With Cannula (N=26) | Delayed-treatment BBL With Cannula (N=21)
Dry eye (Eye disorders) | 1 | 2 | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 3 | 0 | 0
Injection Site Swelling (General disorders) | 4 | 3 | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 6 | 0 | 0 | 0 | 0
Visual acuity tests abnormal (Investigations) | 1 | 4 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT04594239/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT04594239/SAP_001.pdf